CLINICAL TRIAL: NCT00676494
Title: A Prospective, Single Arm, Multi-Center Study to Assess Performance of the Pathway PV Atherectomy System During Percutaneous Peripheral Vascular (PV) Interventions
Brief Title: The Pathway PVD Study for Percutaneous Peripheral Vascular Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pathway Medical Technologies Inc. (Industry)
Responsible Party: Kevin Peters, Director of Clinical Affairs, Pathway Medical Technologies Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC 05003
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Results first posted 2009-07-09 (Estimated); Last update posted 2009-07-09 (Estimated); Status verified 2009-05

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Pathway PV Atherectomy System — The Pathway PV Atherectomy System is a rotating, aspirating, expandable catheter for active removal of atherosclerotic debris and thrombus in lower limb peripheral vasculature during percutaneous interventional procedures.

SUMMARY:
The Pathway PV Atherectomy System is a rotating, aspirating, expandable catheter for active removal of atherosclerotic debris and thrombus in peripheral vasculature.

This is a prospective, single arm, multi-center study to obtain safety and performance data for the Pathway PV Atherectomy System when used as a primary or adjunctive therapy for percutaneous intervention to remove atherosclerotic disease, debris, and thrombus from the lower limb peripheral vasculature.

ELIGIBILITY:
Inclusion Criteria:

* Documented symptomatic atherosclerotic peripheral vascular disease
* Target lesion(s) is/are located in a superficial femoral, popliteal and/or infrapopliteal arteries
* The patient has been informed of the nature of the study and has provided informed consent
* The patient agrees and has capability to meet study requirements and be present at the follow-up clinic visits

Exclusion Criteria:

* Target lesion is located in the iliac artery.
* Target lesion stenosis is < 70%.
* Interventional treatment is intended for in-stent restenosis at the peripheral vascular site.
* Patient is unable to participate for the duration of the study.
* Patient is currently participating or has participated in a study with another investigational medical device or medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2006-02; Primary Completion 2007-07 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Herz Zentrum Bad Krozingen, Germany; Dierk Scheinert, MD, Principal Investigator — University of Leipzig

REFERENCES:
- [Derived] Zeller T, Krankenberg H, Steinkamp H, Rastan A, Sixt S, Schmidt A, Sievert H, Minar E, Bosiers M, Peeters P, Balzer JO, Gray W, Tubler T, Wissgott C, Schwarzwalder U, Scheinert D. One-year outcome of percutaneous rotational atherectomy with aspiration in infrainguinal peripheral arterial occlusive disease: the multicenter pathway PVD trial. J Endovasc Ther. 2009 Dec;16(6):653-62. doi: 10.1583/09-2826.1. PMID 19995118

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: Patients meeting eligibility criteria and enrolled in the study.
Period: Overall Study
Arm/Group | All Patients
Started | 172
Completed | 158
Not Completed | 14
Not completed — Missed Visit | 8
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 134
Age Continuous [Mean (Standard Deviation); unit: years] | 71.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 84
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Secondary Outcome: Average Rutherford Classification Score at 6 Months
Description: Rutherford Classification measures lower limb peripheral arterial disease (PAD) by evaluating and rating symptoms. Score: 0 (no symptoms or discomfort in leg) to 6 (Tissue loss or gangrene in leg)
Time Frame: 6 months
Population: Number of study participants was statistically determined by protocol-defined endpoints. Analysis endpoints were assessed via summary statistics and 95% confidence intervals. No p-values were generated and no statistical inferences asserted regarding point estimates or confidence limits generated for any additional post-hoc data analysis.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | All Patients
Number analyzed (Participants) | 135
Score on scale | 1.5 (1.4)

2. Secondary Outcome: Average Ankle Brachial Index (ABI) at 6 Months
Description: Ankle Brachial Index (ABI) is the ratio of the blood pressure in the lower legs to the blood pressure in the arms. Compared to the arm, lower blood pressure in the leg is a symptom of peripheral artery disease (PAD). Range: Normal arteries (1.0 - 1.2) to Severe arterial disease (under 0.5)
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | All Patients
Number analyzed (Participants) | 138
units on scale | 0.77 (0.26)

3. Secondary Outcome: Freedom From Target Lesion Revascularization (TLR) at 6 Months
Description: Number of patients that did not require target lesion revascularization 6 months after index procedure.
Time Frame: 6 months
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 172
participants | 147

4. Primary Outcome: Major Adverse Events (MAEs) Within 30 Days
Description: Major adverse events (MAEs) are any death, target vessel revascularization (TVR), target lesion revascularization (TLR), myocardial infarction (MI), or amputation of the treated limb that occurred within 30 days of the index procedure.
Time Frame: 30 days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 172
Participants | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators will have the right to publish results of the Study, provided that Investigators submit copies of any proposed publication to Sponsor for review at least 30 days and up to 60 days in advance of publication. Sponsor may extend such review period for another 90 days to file patent applications or protect its Related Rights.